CLINICAL TRIAL: NCT05465928
Title: Neuroimaging Biomarker-Guided Personalized Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment for Major Depressive Episode in Adolescents and Young Adults with Mood Disorders: a Randomized, Double-Blind, Controlled Study
Brief Title: Personalized Repetitive Transcranial Magnetic Stimulation Treatment for Major Depressive Episode
Acronym: PRTMSTMDEAYA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu Province Nanjing Brain Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 81725005-2
Record Dates: First submitted 2022-06-22; First posted 2022-07-20 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-01

CONDITIONS: Major Depressive Episode
Keywords: Repetitive Transcranial Magnetic Stimulation; Major Depressive Episode; Functional Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalized rTMS (Experimental): The active arm will receive the personalized rTMS treatment with parameters as follows:
  1. Neuroimaging biomarker-guided personalized selection for stimulation frequency: low frequency(1HZ) or high frequency (10HZ);
  2. Neuroimaging biomarker-guided personalized selection for stimulation site: dorsalmedial prefrontal cortex or occipital cortex;
  3. Schedule: 2 sessions per day, five days per week for a total of 20 sessions over 2 weeks.
  Interventions: Device: Active rTMS
- sham stimulation rTMS (Sham Comparator): Sham stimulation arm will receive the same scheme of rTMS but with a sham coil.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Active rTMS — rTMS is a non-invasive neuromodulation therapy which has been recognized as a helpful treatment for depression. During each rTMS treatment, the magnetic field is generated by a coil which is placed on the head near the brain region of interest, and further, an electrical current is induced to modulate brain activity.
  Other Names: VISHEE Magneuro stimulator
  Arms: Personalized rTMS
Device: Sham rTMS — The sham rTMS stimulation is performed based on a sham coil which will mimic scalp sensations and the acoustic artifact of the active stimulation, without delivering any magnetic pulse.
  Arms: sham stimulation rTMS

SUMMARY:
Adolescents and young adults with mood disorders experiencing major depressive episode have poor efficacy of medication treatment. Repetitive magnetic transcranial stimulation (rTMS) has been proven adjuvant efficacy in patients with major depressive episode. However, the optimal evidence-based stimulation parameters have not been clearly defined, which greatly limits the efficacy of rTMS in the treatment of major depressive episode.

This trial will compare a novel form of personalized rTMS treatment protocol guided by neuroimaging biomarkers to the sham stimulation.The personalized selection of stimulation parameters, such as stimulation site, frequency and magnetic pulse number, will be determined by neuroimaging biomarkers.

The study aims to propose a novel personalized neuroimaging-guided rTMS strategy, to evaluate the efficacy and safety of the treatment, further to understand the biological mechanism of the personalized rTMS treatment.

DETAILED DESCRIPTION:
Mood disorders, including mainly bipolar disorder (BD) and major depressive disorder (MDD), have become the primary health problem and one of the leading causes of functional disability in adolescents and young adults. In China, the incidence of mood disorders such as BD and MDD in adolescents and young adults has increased rapidly in recent years. Particularly, mood disorder patients currently experiencing major depressive episode are considered to be at high risk for suicide, and pharmacological treatment showed poor efficacy to such depressive patients. Mood disorders with major depressive episode have become one of the main threats to youth mental health in China. Therefore, it is of great significance to explore a series of early intervention strategies for adolescents and young adults with major depressive episode.

rTMS is a non-invasive brain stimulation treatment strategy with mild side effects. In 2008, rTMS was approved by the Food and Drug Administration (FDA) for the treatment of major depression. The selection of stimulation parameters often has a vital impact on the clinical efficacy of rTMS treatment. Several clinical trials have reported the efficacy and safety of rTMS on treatment resistant major depression. However, the evidence-based optimal targets and other stimulation parameters have not been clearly defined, which greatly limits the efficacy of rTMS in the treatment of major depressive episode. To date, there is no large randomized clinical trial (RCT) exploring an optimization of rTMS on adolescents and young adults with major depressive episode.

This study is a double-blind randomized controlled trial aiming at assessing the efficacy and safety of a novel personalized rTMS treatment protocol compared to sham stimulation for major depressive episode in adolescents and young adults with mood disorders. Participants will be assigned randomly (1:1) to the personalized rTMS group or the sham stimulation group. Participants in the rTMS group will be treated with 20 sessions (2 sessions per day) of personalized rTMS treatment, and participants in the sham stimulation group will receive the same scheme of rTMS treatment but with sham coil. The selection of stimulation parameters (stimulation site, frequency, number of pulses, number of sessions, train and inter-train duration) in both groups will be based on neuroimaging biomarkers extracted via machine learning method. Participants in both groups will maintain the stable drug regimen during the rTMS trial.

At baseline and after each 10 sessions of treatment, patients will receive the assessment of depressive symptom severity, cranial magnetic resonance imaging (MRI) scan and peripheral blood collection (about 15ml peripheral blood). Before and after 20 sessions of treatment, neurocognitive function test will be performed. The purposes of the present study are to: 1) evaluate the clinical response to the personalized rTMS treatment by comparing the change in depressive symptom and neurocognitive function over the course of rTMS trial. 2) further understand the possible biological mechanism underlying the efficacy of personalized rTMS treatment by analyzing alterations from multidimensional data of neuroimaging, plasma proteomics and metabolomics.

ELIGIBILITY:
Inclusion Criteria:

* Between 13 and 25 years of age;
* Participants fulfill the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnostic criteria for major depressive disorder (MDD) or bipolar disorder (BD). Participants are assessed by the Structured Clinical Interview for DSM-IV for Axis I Disorders (SCID-I, patients' age ≥18 years old), or the Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime version (K- SADS-PL, patients' age< 18 years old);
* A current moderate or severe depressive episode defined by HAMD≥17 and Young Mania Rating Scale (YMRS) <12;
* Participants receive a stable psychotropic medication regimen prior to randomization to the trial and are willing to remain on the stable regimen during the rTMS treatment phase;
* Participants and 1 or 2 parents (patients' age< 18 years old) provide informed consent after the detailed description of the study.

Exclusion Criteria:

* Prior rTMS or electroconvulsive therapy (ECT) treatment or standard psychological therapy within 6 months prior to screening;
* Comorbidity of other DSM-IV axis I disorders or personality disorders;
* Judged clinically to be at serious suicidal risk;
* Diabetes mellitus, hypertension, vascular and infectious diseases and other major medical comorbidities;
* Unstable medical conditions, e.g., severe asthma;
* Neurological disorders, e.g., history of head injury with loss of consciousness for ≥ five minutes, cerebrovascular diseases, brain tumors and neurodegenerative diseases;
* Mental retardation or autism spectrum disorder;
* Contraindications to MRI (e.g., severe claustrophobia, pacemakers, metal implants);
* Contraindications to rTMS (e.g., metal in head, history of seizure, electroencephalogram (EEG) test suggesting high risk of seizure, known brain lesion);
* Current drug/alcohol abuse or dependence;
* Pregnant or lactating female.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 219 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in depressive symptoms assessed by Hamilton depression rating scale 17 items (HAMD-17) at week 1 and week 2. | Baseline, week 1 and week 2.
  The HAMD-17 scale has 17 items. The total score ranges from 0-52, with higher score indicating more severe depressive symptoms. A total score of 0-7 is considered to be normal. Scores of 17 or higher indicate moderate, severe, or very severe depression.
Change from baseline in the amplitude of low-frequency fluctuation (ALFF) values measured by resting-state functional magnetic resonance imaging (fMRI) at week 1 and week 2. | Baseline, week 1 and week 2.
  Participants will undergo fMRI scans prior to beginning rTMS treatment (week 0) and after completing 10 sessions of rTMS treatment (weeks 1) and after completing 20 sessions of rTMS treatment (weeks 2). ALFF is a fMRI indicator that reflects the spontaneous neural activity. After data acquisition, whole-brain voxel-wise analysis of ALFF values will be performed to detect the change from baseline in brain functional activity at week 1 and week 2.
Change from baseline in neurocognitive function using Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) test at week 2. | Baseline and week 2.
  RBANS is a test for identifying and characterizing abnormal cognitive decline for patients with neuropsychiatric disorders. The RBANS is comprised of five domains, which are Immediate Memory, Visuospatial /Constructional, Language, Attention and Delayed Memory. The total score of RBANS range from 40-160, with 160 referring to higher cognitive functioning. A score of 95-115 is in the average range; score of 70-85 mild to moderate cognitive impairment; score <70 moderate to severe impairment.

SECONDARY OUTCOMES:
Change from baseline in the Clinical Global Impression-Severity scale (CGI-S) at week 1 and week 2. | Baseline, week 1 and week 2.
  The CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. A rating of 1 is considered normal, or with the least severe symptoms, a rating of 7 is extremely ill, or the worst symptoms.
Change from baseline in the Montgomery-Asberg Depression Rating Scale (MADRS) at week 1 and week 2. | Baseline, week 1 and week 2.
  MADRS is a clinician-rated scale used to assess depressive symptom severity and detect changes due to antidepressant treatment. The scale consists of 10 items, each of which is rated from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms). The total score of MADRS ranges from 0 to 60, with higher score indicating more severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Wang, Study Chair — Affiliated Nanjing Brain Hospital, Nanjing Medical University
Locations (1):
- Affiliated Nanjing Brain Hospital, Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalin NH. Advances in Understanding and Treating Mood Disorders. Am J Psychiatry. 2020 Aug 1;177(8):647-650. doi: 10.1176/appi.ajp.2020.20060877. No abstract available. PMID 32741277
- [Background] Nesvag R, Bramness JG, Handal M, Hartz I, Hjellvik V, Skurtveit S. The incidence, psychiatric co-morbidity and pharmacological treatment of severe mental disorders in children and adolescents. Eur Psychiatry. 2018 Mar;49:16-22. doi: 10.1016/j.eurpsy.2017.12.009. Epub 2018 Feb 3. PMID 29366845
- [Background] Rumi DO, Gattaz WF, Rigonatti SP, Rosa MA, Fregni F, Rosa MO, Mansur C, Myczkowski ML, Moreno RA, Marcolin MA. Transcranial magnetic stimulation accelerates the antidepressant effect of amitriptyline in severe depression: a double-blind placebo-controlled study. Biol Psychiatry. 2005 Jan 15;57(2):162-6. doi: 10.1016/j.biopsych.2004.10.029. PMID 15652875
- [Background] Rosenich E, Gill S, Clarke P, Paterson T, Hahn L, Galletly C. Does rTMS reduce depressive symptoms in young people who have not responded to antidepressants? Early Interv Psychiatry. 2019 Oct;13(5):1129-1135. doi: 10.1111/eip.12743. Epub 2018 Oct 10. PMID 30303308
- [Background] Mayer G, Aviram S, Walter G, Levkovitz Y, Bloch Y. Long-term follow-up of adolescents with resistant depression treated with repetitive transcranial magnetic stimulation. J ECT. 2012 Jun;28(2):84-6. doi: 10.1097/YCT.0b013e318238f01a. PMID 22531199
- [Background] Hett D, Rogers J, Humpston C, Marwaha S. Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Depression in Adolescence: A Systematic Review. J Affect Disord. 2021 Jan 1;278:460-469. doi: 10.1016/j.jad.2020.09.058. Epub 2020 Sep 15. PMID 33011525
- [Background] Weigand A, Horn A, Caballero R, Cooke D, Stern AP, Taylor SF, Press D, Pascual-Leone A, Fox MD. Prospective Validation That Subgenual Connectivity Predicts Antidepressant Efficacy of Transcranial Magnetic Stimulation Sites. Biol Psychiatry. 2018 Jul 1;84(1):28-37. doi: 10.1016/j.biopsych.2017.10.028. Epub 2017 Nov 10. PMID 29274805
- [Background] Fox MD, Buckner RL, White MP, Greicius MD, Pascual-Leone A. Efficacy of transcranial magnetic stimulation targets for depression is related to intrinsic functional connectivity with the subgenual cingulate. Biol Psychiatry. 2012 Oct 1;72(7):595-603. doi: 10.1016/j.biopsych.2012.04.028. Epub 2012 Jun 1. PMID 22658708
- [Background] Downar J, Geraci J, Salomons TV, Dunlop K, Wheeler S, McAndrews MP, Bakker N, Blumberger DM, Daskalakis ZJ, Kennedy SH, Flint AJ, Giacobbe P. Anhedonia and reward-circuit connectivity distinguish nonresponders from responders to dorsomedial prefrontal repetitive transcranial magnetic stimulation in major depression. Biol Psychiatry. 2014 Aug 1;76(3):176-85. doi: 10.1016/j.biopsych.2013.10.026. Epub 2013 Nov 28. PMID 24388670
- [Background] Chang M, Womer FY, Gong X, Chen X, Tang L, Feng R, Dong S, Duan J, Chen Y, Zhang R, Wang Y, Ren S, Wang Y, Kang J, Yin Z, Wei Y, Wei S, Jiang X, Xu K, Cao B, Zhang Y, Zhang W, Tang Y, Zhang X, Wang F. Identifying and validating subtypes within major psychiatric disorders based on frontal-posterior functional imbalance via deep learning. Mol Psychiatry. 2021 Jul;26(7):2991-3002. doi: 10.1038/s41380-020-00892-3. Epub 2020 Oct 1. PMID 33005028
- See also: Depression — http://www.who.int/mediacentre/factsheets/fs369/en/.